CLINICAL TRIAL: NCT03339622
Title: Safety and Efficacy of PPP001-kit for Improving Health Related Quality of Life in Advanced Cancer Patients With Uncontrolled Pain: A Randomized, Double-blind, Placebo-Controlled, Parallel Group Study
Brief Title: Safety and Efficacy of Smoked Cannabis for Improving Quality of Life in Advanced Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Mycotoxin potential contamination of one lot of study drug
Sponsor: Tetra Bio-Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPP001-Ph3-01
Record Dates: First submitted 2017-10-17; First posted 2017-11-13 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Cancer; Chronic Pain Due to Malignancy (Finding)
Keywords: uncontrollable cancer pain; incurable malignancy,
MeSH Terms: conditions — Neoplasms; Signs and Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smoked cannabis (PPP001) (Experimental): 280 mg dried cannabis pellet -(9% THC / 2% CBD per pellet)
  Interventions: Combination Product: PPP001
- THC free placebo (Placebo Comparator): 280 mg dried extracted cannabis pellet (0% THC / 0.6% CBD per pellet)
  Interventions: Combination Product: placebo

INTERVENTIONS:
Combination Product: PPP001 — 1 pellet smoked three times a day with titanium pipe (280 mg dried cannabis pellet - 9% THC / 2% CBD per pellet)
  Other Names: titanium pipe
  Arms: smoked cannabis (PPP001)
Combination Product: placebo — 1 pellet smoked three times a day with titanium pipe (280 mg dried cannabis pellet - 0% THC / 0.6% CBD per pellet)
  Other Names: titanium pipe
  Arms: THC free placebo

SUMMARY:
Cancer causes pain in many of the patients that it affects. Physicians specialized in palliative care help advanced cancer patients to maintain as good pain control as possible through the use of medications such as opioids. Even with palliative care and optimal use of medications, many patients still suffer enormously as the cancer spreads. Because of this, some cancer patients also try or use cannabis in different ways to relieve their pain and improve the way they feel. However, there has not been much high-quality research done yet to prove whether or not cannabis products are truly useful to relieve severe cancer pain. This study is to test if advanced cancer patients who use inhaled medical cannabis (PPP001), in addition to palliative care management, will experience improvement in quality of life and relieve uncontrolled pain, providing safety conditions.

DETAILED DESCRIPTION:
This is a 4-week randomized, double-blind, placebo-controlled, parallel group design trial to evaluate the safety and efficacy of inhaled PPP001 to improve quality of life (HRQoL) and reduce pain intensity, in patients with uncontrolled cancer pain and incurable malignancy.

Nine hundred forty six adult patients, male and female, with chronic cancer pain (at least 3 months in duration) and advanced disease, with an average weekly pain intensity score greater than 4 on a 11 points Numerical Rate Scale (NRS), will be prospectively recruited and invited to participate in this trial.

Informed consent will be obtained by a Research Assistant.

After baseline documentation with standardized scales, patients will be randomized to one of 2 parallel groups:

Group A: 4 weeks PPP001-kit three times daily; Group B: 4 weeks placebo-kit three times daily; The inhalation of PPP001 or placebo-kit will be allowed three times a day at 4-6 hour intervals. Rescue medication will also be allowed.

Patients will have a dose titration phase during the first week, followed by an additional 3-week period of treatment. The dose escalation will allow patients to adapt to the potential AEs of cannabis.

Patients will have follow-up after 1 week and 4 weeks of treatment. Once the patient has completed 4 weeks of inhaled PPP001 or placebo, it will be rolled into a long-term follow-up phase until drop-out or death. All patients, including the ones in the placebo group, will be allowed to receive the active treatment once the 4-weeks trial has finished, and continue it until death or drop-out.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Adult male and female patients at least 18 years of age
3. Subject agreed to follow the protocol
4. Advanced cancer for which there is no known curative therapy
5. Patients experiencing pain ≥4 on NRS due to cancer related pain
6. Life expectancy six weeks or longer
7. PPI score less than or equal to 4 (survival more than 6 weeks)
8. PPS greater than or equal 70%
9. PaP Score Group A (30-day survival probability >70%)
10. An Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
11. The patient has a clinical diagnosis of cancer related pain, which is not alleviated with their current optimized opioid treatment
12. The patient is using no more than one type of breakthrough opioid analgesia
13. Normal cognitive status according to MDAS and MiniCog
14. Normal liver function (defined as aspartate aminotransferase 10-40 U/L and alanine aminotransferase 7-56 U/L)
15. Normal renal function (defined as serum creatinine level <133 µmol/L and Estimated Glomerular Filtration Rate (eGFR) greater than or equal to 60)
16. The patient is able to perform deep inhalations and hold breath for at least 5 to 10 seconds. If there is any pulmonary disease diagnosed previously (obstructive and/or restrictive pathology), the patient must be able to perform a maximal inhalation of at least 12-15 ml/kg measured with an incentive spirometer, followed by a normal exhalation
17. Ability to read and respond to questions in French or English.
18. Previous or current use of opioid analgesics (at least 1 week)
19. A female volunteer must meet one of the following criteria:

    If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first drug administration, during the study and for at least 60 days after the last dose. An acceptable method of contraception includes one of the following:
    * Abstinence from heterosexual intercourse
    * Systemic contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
    * Intrauterine device (with or without hormones)
    * Condom with spermicide or condom with intravaginally applied spermicide If of non-childbearing potential - should be surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least one year without menses)
20. A male volunteer with sexual partners who are pregnant, possibly pregnant, or who could become pregnant must meet the following criteria:

    * Participant is unable to procreate, defined as surgically sterile (i.e. has undergone a vasectomy within the last 6 months)
    * Participant agrees to use one of the accepted contraceptive regimens from first drug administration until 3 months after the last drug administration. An acceptable method of contraception includes one of the following:

A. Abstinence from heterosexual intercourse. B. Condom with spermicide or condom with intravaginally applied spermicide

Exclusion Criteria:

1. Pain due to other causes different than cancer related pain
2. Previous serious adverse event or hypersensitivity to cannabis or cannabinoids
3. Inability to understand and comply with the instructions of the study
4. Presence of significant cardiac disease (history of unstable ischemic heart disease, heart failure, severe and uncontrolled hypertension) that, in the opinion of the investigator, would put the patient at risk of a clinically significant arrhythmia or myocardial infarction
5. Current substance use disorder according to the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM 5)
6. Life-time history of dependence on cannabis or diagnosis of cannabis use disorder (CUD) according to the DSM 5
7. Life-time history of DSM 5 schizophrenia, bipolar disorder, or previous psychosis with or intolerance to cannabinoids
8. Current or history of suicidal ideation according to the Columbia-Suicide Severity Rating Scale (C-SSRS) approved by FDA in 2012 for assessment of suicidal ideation and behaviour
9. Pregnant, breast-feeding or female patients of child-bearing potential and male patients whose partner is of child-bearing potential, unless willing to ensure that they or their partner use effective contraception, for example, oral contraception, double barrier, intra-uterine device, during the study and for three months thereafter (however, a male condom should not be used in conjunction with a female condom as this may not prove effective)
10. Hepatic impairment (aspartate aminotransferase more than three times normal) or renal function impairment (serum creatinine level >133 µmol/L, Estimated Glomerular Filtration Rate (eGFR) <60)
11. Cognitive impairment according to MDAS and MiniCog
12. Patient has any planned clinical interventions that would affect their pain (e.g., chemotherapy or radiation therapy where, in the clinical judgment of the investigator, these would be expected to affect pain)
13. Cancer treatments that may interfere with stability of treatment (epidural, radiotherapy, chemotherapy, hormonal therapy)
14. Epilepsy
15. The patient is currently using or has used cannabinoid based medications within 30 days of study entry and is unwilling to abstain for the duration of the study
16. Positive urine drug screen for cannabinoids and other potential abuse substances (e.g. alcohol, cocaine, amphetamines and methamphetamines, hallucinogens, unprescribed opioids and ketamine, etc.)
17. Participation in another clinical trial within 30 days of enrolment in our trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
improve Health Related Quality of Life (HRQoL) of patients with uncontrolled cancer pain and incurable malignancy | Change from Baseline in HRQoL at Weeks 1 and 4. Change from baseline at 12-weeks follow-up and every 6-weeks after week 12 follow-up until the date of death from any cause or assessed up to 12 months.
  Does the daily use of PPP001-kit improve European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 15 Palliative (EORTC-QLQ-C15-PAL). Scale range is 1 to 4; 1 (Not at All) being the worst rating to the maximal rating of 4 (Very Much).

SECONDARY OUTCOMES:
Does the daily use of PPP001-kit improve uncontrolled cancer pain | Change from Baseline in BPI-SF at Weeks 1 and 4. Change from baseline at 12-weeks follow-up and every 6-weeks after week 12 follow-up until the date of death from any cause or assessed up to 12 months
  Changes in pain as measured by the Brief Pain Inventory-Short Form (BPI-SF) scale. Scale range is 0 to 10; 0 (No pain) being the best rating to the maximal rating of 10 (Pain as bad as you can imagine).
Does the daily use of PPP001-kit improve symptom burden | Change from Baseline in ESAS-r-CS at Weeks 1 and 4. Change from baseline at 12-weeks follow-up and every 6-weeks after week 12 follow-up until the date of death from any cause or assessed up to 12 months
  Changes in symptom burden as measured by the revised Edmonton Symptom Assessment System version with Constipation and Sleep was added to assess improvement in symptom burden (ESAS-r-CS). Scale range is 0 to 10; 0 (No symptom) being the best rating to the maximal rating of 10 (Worst possible score for symptom).
Does the daily use of PPP001-kit improve functional status | Change from Baseline in PPSv2 at Weeks 1 and 4. Change from baseline at 12-weeks follow-up and every 6-weeks after week 12 follow-up until the date of death from any cause or assessed up to 12 months
  Changes in Palliative Performance Scale (PPSv2) version 2. Scale range is a left to right and downward scale for participant to find the best description of their palliative performance. Worst being 0% score representing Dead to PPS 100% representing Full ability to interact and function.
Does the daily use of PPP001-kit improve the QoL of family caregivers | Change from Baseline in CQOLC at Weeks 1 and 4
  Changes in Caregivers Quality of Life Index- Cancer (CQOLC). Scale range is 0 to 4; 0 meaning Not at All affected and 4 meaning Very Much affected.
Changes in validated Udvalg for klinische Undersøgelser (UKU) Side Effects Rating Scale, Self-rating version for Patients (UKU-SERS-Pat) | Change versus placebo for safety and tolerability at Weeks 1 and 4. Change from baseline at 12-weeks follow-up and every 6-weeks after week 12 follow-up until the date of death from any cause or assessed up to 12 months.
  Changes in validated Udvalg for klinische Undersøgelser (UKU) Side Effects Rating Scale, Self-rating version for Patients (UKU-SERS-Pat). Scale range is 0 to 3 for rating the degree of severity and a second scale for the investigator that assigns a casual relationship of improbable, possible or probable.
Does the daily use of PPP001-kit improve cognition | Change versus placebo for Mini-Cog at Weeks 1 and 4. Change from baseline at 12-weeks follow-up and every 6-weeks after week 12 follow-up until the date of death from any cause or assessed up to 12 months
  Changes in validated Mini-Cog. Scale range is numerical and rates the ability to recall words and ability to draw a clock showing numbers from 1 to 12 and then drawing the given time.
Does the daily use of PPP001-kit influence pharmacodynamics | Change versus placebo for 100-mm VAS at Weeks 1 and 4
  Changes in a 100-mm VAS of good drug effect, and a VAS for the items "high," "relaxed," "stressed," and "happy" (0 = not at all, 10 = extremely)
Does the daily use of PPP001-kit influence the use of concurrent medications | Change from Baseline in MQS version III at Weeks 1 and 4.
  Changes in concurrent medications will be measured using the Medication Quantification Scale (MQS) version III. The MQS version III is a method of quantifying different pain drug regimens by evaluating the use of 22 distinct drug classes (e.g., nonsteroidal anti-inflammatory drugs [NSAIDs], antidepressants, benzodiazepines, opiates). A single value is calculated based on a patient's pain medication profile, taking into account dosages, and the types of pain medications prescribed.
Does the daily use of PPP001-kit improve quality of life | Change from Baseline in EQ-5D at Weeks 1 and 4. Change from baseline at 12-weeks follow-up and every 6-weeks after week 12 follow-up until the date of death from any cause or assessed up to 12 months
  Changes in validated European Quality of Life-5 Dimensions (EQ-5D). First scale range provides 5 statements that describe the participants health TODAY; it includes 5 different health assessments. The second scale is 0 to 100 and requires that the participant places a mark on the scale showing how good or bad they feel TODAY; 0 meaning The worst health they can imagine; 100 meaning the best health they can imagine.
Does the daily use of PPP001-kit improve uncontrolled cancer pain | Change from Baseline in NRS at Weeks 1 and 4. Change from baseline at 12-weeks follow-up and every 6-weeks after week 12 follow-up until the date of death from any cause or assessed up to 12 months
  Changes in pain as measured by the Numerical Rating Scale (NRS). The NRS is a measure of the average weekly pain intensity score greater than on a 0 to 10 points scale where 0 is No Pain and 10 is the worst pain.
Does the daily use of PPP001-kit improve mood and illness-understanding | Change versus placebo for MDAS at Weeks 1 and 4. Change from baseline at 12-weeks follow-up and every 6-weeks after week 12 follow-up until the date of death from any cause or assessed up to 12 months
  Changes in validated Memorial Delirium Assessment Scale (MDAS). Scale range is 0 to 3; 0 meaning None and 3 meaning Severe.
Does the daily use of PPP001-kit influence the use of the need for rescue medication | Change from Baseline in rescue medication reported as an MEDD at Weeks 1 and 4.
  Rescue medication will be based on the calculation of 10% of the total morphine equivalent daily dose (MEDD). The reduction or increase in the total MEDD will be recorded after starting treatment with PPP001.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Vigano, MD, MSc, Principal Investigator — McGill University
Locations (1):
- Sante Cannabis, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided